CLINICAL TRIAL: NCT05508152
Title: Prophylaxis of Surgical Wound Infection in Incisional Hernia Repair With Topical Antibiotics (PROTOP-PAR)
Acronym: (PROTOP-PAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PROTOP-PAR
Record Dates: First submitted 2022-05-04; First posted 2022-08-19 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Hernia
Keywords: Surgical site infection; Incisional hernia; Topical prophylaxis; Wound irrigation; Topical antibiotic prophylaxis
MeSH Terms: conditions — Incisional Hernia; Surgical Wound Infection | interventions — Amoxicillin-Potassium Clavulanate Combination; Saline Solution; Anti-Bacterial Agents; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound irrigation with saline (Sham Comparator): After the closure of the aponeurosis, and before the closure of the skin, the subcutaneous layer of the wound will be rinsed with a determined volume (depending on the diameter of the incision) of a saline solution. Then, a gauze soaked with the same solution will be placed in the wound for 3 minutes.
  Interventions: Drug: Wound irrigation with a saline solution
- Wound irrigation with antibiotic (Experimental): After the closure of the aponeurosis, and before the closure of the skin, the subcutaneous layer of the wound will be rinsed with a determined volume (depending on the diameter of the incision) of amoxicillin-clavulanate in saline solution. Then, a gauze soaked with the same solution will be placed in the wound for 3 minutes.
  Interventions: Drug: Wound irrigation with amoxicillin-clavulanate in saline solution

INTERVENTIONS:
Drug: Wound irrigation with amoxicillin-clavulanate in saline solution — Randomization will be made by means of the RedCap online program. At the arrival of the patient in the surgical area, the nursing team will be informed whether or not the patient has entered the protocol of the studio.
  For each included case, the perioperative nurse will access RedCap and will proceed to include and randomize the case.
  Once the patient's data has been introduced, the circulating nurse will enter the intervention group in a registration database, keeping it blinded to the surgical team.
  In the experimental arm of the study, the circulating nurse will prepare a solution of amoxicillin-clavulanate acid (1000 mg of antibiotic in 500 mL of saline) outside the operating room. In case of open surgery, the thickness of the subcutaneous fat layer will be measured and recorded. After the closure of the aponeurosis, and before the closure of the skin, the wound will be irrigated with the antibiotic solution, and the soaked gauze placed on the wound for 3 minutes.
  Other Names: Antibiotic
  Arms: Wound irrigation with antibiotic
Drug: Wound irrigation with a saline solution — Randomization will be made by means of the RedCap online program. At the arrival of the patient in the surgical area, the nursing team will be informed whether or not the patient has entered the protocol of the studio. For each included case, the perioperative nurse will access RedCap and will proceed to include and randomize the case.
  Once the patient's data has been introduced, the circulating nurse will enter the intervention group in a registration database, keeping it blinded to the surgical team.
  If the case belongs to the sham group, at the end of the intervention, the circulating nurse will prepare a sham solution contaning only normal saline outside the operating room. In case of open surgery, the thickness of the subcutaneous fat layer will be measured and recorded. After the closure of the aponeurosis, and before the closure of the skin, the wound will be irrigated with saline, and the soaked gauze placed on the wound for 3 minutes.
  Other Names: Saline
  Arms: Wound irrigation with saline

SUMMARY:
Surgical site infection (SSI) is the main complication of surgery. The prevention of superficial SSI by topical prophylaxis is controversial. Human studies on wound lavage with topical solutions (saline, antiseptics or antibiotics) are old and do not yield conclusive results. In experimental conditions there is evidence in favor of the efficiency wound lavage with saline and antibiotic solutions. Clinical studies are needed to demonstrate the safety and efficacy of antibiotic lavage.

Objective. Study of the efficacy of topical antibiotic therapy in the prevention of SSI in patients undergoing incisional hernia repair after abdominal surgery.

Method. Randomized double-blind clinical trial comparing two groups of topical prophylaxis. Follow-up will be 90 days after operation. Data will be collected anonymously and the relationships between the variables will be analyzed using Pearson's chi-square, survival analysis and analysis of risk factors as appropriate. The effect of topical antibiotic on hospital stay, resistance patterns in SSI, and antibiotic serum levels will be analyzed.

DETAILED DESCRIPTION:
Several Surgical site infection (SSI) prevention guidelines have been published over the last 10 years. Topical prophylaxis of the surgical wound with antibiotics or antiseptics is one of the most controversial measures proposed for SSI prevention. Two guidelines (British, Spanish Ministry of Health) explicitly recommend not irrigating surgical wounds with any product. The World Health Organization considers irrigation with antibiotics as an unresolved issue and, together with the Centers for Disease Control, recommends irrigation with a solution of povidone iodine. The other four guides do not mention the measure. In Catalonia, a SSI prevention bundle recommends wound irrigation with saline, with a low level of recommendation.

Therefore, topical prophylaxis with operational wound washings with different solutions has been poorly studied, evokes contradictory recommendations and is not included in the majority of clinical practice guidelines for SSI prevention.

However, a high level of use of wound irrigation at the end of an intervention in actual clinical practice has been observed. In a survey conducted by 2017 and answered by 845 general surgeons of the Spanish Association of Surgeons, before closing the skin, most surgeons (80.6%) irrigate the subcutaneous layer of the wound, either with saline (51.2%), an antiseptic solution (23.8%) or an antibiotic solution (1.5%). Only 19.4% of respondents do not irrigate. In another survey in 2018, focused on colorectal surgeons of two Spanish associations, similar rates of irrigation with saline, antiseptic or antibiotic were used (55%, 28.9% and 2.2%, respectively).

SSI rates after complex incisional hernia repair are higher than previously reported. In a recent paper, this research team observed that patients with SSI after hernia repair showed more prolonged surgical procedures, and a higher one-year recurrence rate. Multivariable analysis revealed the only identified risk factor for SSI to be post-operative sero-hematomas. Patients who developed an SSI required antibiotic agents and daily treatment from one to five months. One of these required the removal of the mesh. SSI rates were high for incisional hernia surgery (16%), and were associated with local complications.

The hypothesis of the study is that topical prophylaxis of the surgical wound with irrigation with an antibiotic solution decreases the rate of postoperative infection in patients undergoing incisional hernia surgery with different levels of contamination.

The study will compare the efficacy of topical prophylaxis with saline with a solution of amoxicillin-clavulanate in the incidence of SSI in incisional hernia repair.

It is a randomized, controlled, multicenter, blind study by observer and patient, with two parallel study groups, phase IV.

Design of study The irrigation of the wound with 0.9% saline will be compared with the irrigation with an active principle solution of a pharmaceutical specialty of proven efficacy (amoxicillin-clavulanate) by parenteral route, administered topically and dissolved in saline.

The two groups of the study will be named: Study Group (irrigation with antibiotic solution) and Control Group (irrigation with saline).

The project has received the Spanish Drug Agency authorization as a low intervention study, a grant from the Spanish Ministry of Health and the Ethics Committee authorization of the Hospital General of Granollers.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require an elective surgical procedure due to an abdominal wall incisional hernia.

Exclusion Criteria:

* Emergency surgery
* Parastomal hernia
* Patients under treatment with immunosuppressants, corticosteroids and patients on hemodialysis.
* Patients with liver cirrhosis.
* Patients with suspected allergy to bata-lactams antibiotics.
* Patients who have undergone a recent open abdomen surgical technique (up to 30 days pre-intervention), placement of a prosthesis made of synthetic material (mesh) or in which the wound cannot be closed surgery at the discretion of the surgeon.
* Patients defined as grade 5 of the American Association of Anaesthesiologists classification (ASA 5).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection rate | 90 days
  The primary study end point will be the development of a Surgical Site Infection (SSI) within 90 days of operation, according to the definitions of the Centres for Disease Control and Prevention (CDC).
  SSI will be defined as superficial incisional (S-SSI), deep incisional (D-SSI) or organ-space (O/S-SSI).
  The incidence of SSI will be measured as events per 100 included procedures.

SECONDARY OUTCOMES:
Hospital stay | 90 days
  To study the effect of topical antibiotic prophylaxis on hospital stay.
Healthcare cost | 90 days
  To study the effect of topical antibiotic prophylaxis on healthcare costs. Using the existing computer systems in the participating hospitals, hospital analytical accounting tools will be used to compare the costs of healthcare between the two groups. Among other items, the costs for hospital stay, surgical interventions, drugs (especially the use of antibiotics), readmissions, medical supplies and staff costs will be analysed.
Bacterial resistance | 90 days
  To analyze the effect of topical antibiotic prophylaxis on the resistance patterns of the flora causing SSI. The percentages of multiresistant bacteria will be compared in the year prior to the start of the study against the period of development of the study in the clinical services participating in the trial. In addition, if there are postoperative infections with positive microbiology results, the percentage of multiresistant bacteria in the sham group will be compared with the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be provided at request